CLINICAL TRIAL: NCT02288260
Title: RuSsian RegisTry of Acute CoronaRy SyndromE TreAtMent and Approach in Dual Antiplatelet Therapy (STREAM)
Brief Title: RuSsian RegisTry of Acute CoronaRy SyndromE TreAtMent and Approach in Dual Antiplatelet Therapy
Acronym: STREAM
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00242
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Russian ACS Registry; ticagrelor
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part A: PATIENTS RECEIVED THE STANDARD MEDICAL CARE AS DETERMINED BY THE TREATING CARDIOLOGIST
- Part B: Patients on ticagrelor at the time of discharge from hospital

SUMMARY:
This NIS is a multi-centre, observational, descriptive, cross-sectional study including all consecutive patients with Acute Coronary Syndrome (ACS) and a single-arm, prospective, longitudinal cohort study which will include patients hospitalized for ACS and who are with ticagrelor on discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Part A,B: Subjects whose data have been entered in the Russian ACS Registry
* PART A,B: Discharged from hospital after MI with ST-segment elevation (STEMI), MI NST segment elevation (NSTEMI) or Unstable angina. Hospitalized during 24 hours of ACS symptoms onset
* Part B: Patients on ticagrelor at the time of discharge from hospital

Exclusion Criteria:

* The existence of serious / severe concomitant diseases which can in the short term (i.e. within 6 months) limit the duration of life
* Current participation in a clinical trial with a non-licensed investigational medicinal product

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study includes patients, in a real-life setting, who are hospitalized for acute coronary syndrome (ACS) within 24 hours of symptom onset and who have a final diagnosis of Unstable Angina (UA), Myocardial Infarction (MI) and were discharged. Including transferred to another medical institution after 24 hours from the moment of hospitalization; transferred from other medical institutions within 24 hours from the moment of initial hospitalization to hospital.
  Principal of choice in the Single-cohort study: only patients with ticagrelor at discharged.
  Patients received the standard medical care as determined by the treating cardiologist.
Sampling Method: Non-Probability Sample
Enrollment: 5470 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving different types of short-term antithrombotic treatment according to different type of acute coronary syndrome (STEMI - ST-elevation myocardial infarction, NSTE(Non-ST-elevation)-ACS and Unstable Angina). (Part A) | 1st Jan of 2012-1st March of 2015
  Patients included in Federal ACS Registry from 1st Jan of 2012 till 1st March of 2015
Proportion of patients taking ticagrelor with cardiovascular (CV) events after discharge from hospital depending on DAT (Dual Antiplatelet Therapy) duration. (Part B) | Up to 2 years
  During follow up

SECONDARY OUTCOMES:
Proportion of patients who undergo invasive or non-invasive short-term clinical management according to different type of acute coronary syndrome (STEMI, NSTE-ACS and Unstable Angina). (Part A) | 1st Jan of 2012-1st March of 2015
  Patients included in Federal ACS Registry from 1st Jan of 2012 till 1st March of 2015
Time from first symptoms onset to the time of hospitalization (Part A) | 1st Jan of 2012-1st March of 2015
  Patients included in Federal ACS Registry from 1st Jan of 2012 till 1st March of 2015
Proportion of patients receiving different types of ACS treatment depending on ACS symptoms duration prior hospitalization. (Part A) | 1st Jan of 2012-1st March of 2015
  Patients included in Federal ACS Registry from 1st Jan of 2012 till 1st March of 2015
Patients demographic and baseline characteristics (age, gender, weight, height). (Part A) | 1st Jan of 2012-1st March of 2015
  Patients included in Federal ACS Registry from 1st Jan of 2012 till 1st March of 2015
Proportion of patients with different type of coronary intervention strategies. (Part A) | 1st Jan of 2012-1st March of 2015
  Patients included in Federal ACS Registry from 1st Jan of 2012 till 1st March of 2015
Proportion of patients who is on ticagrelor treatment during 0-3 months, >3-6 months, >6-9 months, >9-12 months. (Part B) | Up to 2 years
  During follow up
Proportion of patients with ticagrelor treatment interruptions according to different clinical and non-clinical events (bleeds, planned and non-planned medical interventions, etc.) during follow-up. (Part B) | Up to 2 years
  During follow-up period
Proportion of patients with thrombo-embolic events during follow-up depending on DAT therapy duration. (Part B) | Up to 2 years
  During follow-up period
Proportion of patients who discontinued ticagrelor and reason to discontinue ticagrelor treatment. (Part B) | Up to 2 years
  during follow-up period
Proportion of patients with significant violations of treatment regimen with ticagrelor. (Part B) | Up to 2 years
  during follow-up period
Start and stop dates of dual antipatelet therapy and ticagrelor (as part of DAT) and duration of exposure to DAT and ticagrelor in real-life setting. (Part B) | Up to 2 years
  during follow-up period
Proportion of patients who discontinued DAT and the reason of discontinuation of DAT in real-life setting. (Part B) | Up to 2 years
  during follow-up period
Proportion of patients who change DAT components and reason to change of DAT. (Part B) | Up to 2 years
  during follow-up period
Proportion of patients with CV-events (recurrent Myocardial Infarction-MI, stroke, ischemia-driven revascularization, death, etc.) in long-term perspective (second year) after index event in real-life setting. (Part B) | Up to 2 years
  during follow-up period
Proportion of patients using different type of antithrombotic therapy in long-term perspective (second year) after index event. (Part B) | Up to 2 years
  during follow-up period
Proportion of patients who managed by cardiologist, therapist and other physician after discharge from the hospital. (Part B) | Up to 2 years
  during follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Bulatov, MCMD, Study Director — AstraZeneca; Eleva Oschepkova, MD, PROFESSOR OF CARDIOLOGY, Principal Investigator — Russian Cardiology Research and Production Complex
Locations (15):
- Russia (15):
  - Research Site, Arkhangelsk
  - Research Site, Cheboksary
  - Research Site, Irkutsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Petrozavodsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Stavropol
  - Research Site, Tomsk
  - Research Site, Tyumen
  - Research Site, Ufa
  - Research Site, Vladivostok

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00242&attachmentIdentifier=d30a1cc5-a881-45ad-bff9-257f00249024&fileName=D1843R00242_Study_report_synopsis.pdf&versionIdentifier=